CLINICAL TRIAL: NCT02682784
Title: Neural Substrates of Emotion: Impact of Cocaine Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO39699
Record Dates: First submitted 2016-02-08; First posted 2016-02-15 (Estimated); Results first posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-09

CONDITIONS: Cocaine Use Disorder
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Oxytocin/Cocaine User (Experimental): Individuals who meet criteria for cocaine use disorder and are randomized to oxytocin.
  Interventions: Drug: Oxytocin
- Placebo/Cocaine User (Active Comparator): Individuals who meet criteria for cocaine use disorder and are randomized to placebo.
  Interventions: Drug: Placebo
- Oxytocin/Control (Experimental): Healthy controls who are randomized to oxytocin.
  Interventions: Drug: Oxytocin
- Placebo/Control (Active Comparator): Healthy controls who are randomized to placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Nasal spray based on naturally occurring hormone, oxytocin.
  Other Names: Pitocin
  Arms: Oxytocin/Cocaine User; Oxytocin/Control
Drug: Placebo
  Arms: Placebo/Cocaine User; Placebo/Control

SUMMARY:
Over one million individuals in the United States meet criteria for cocaine use disorders. Relapse rates are highest among cocaine-dependent (CD) populations. Social stress is a significant risk factor for relapse. Data from human neuroimaging studies suggest that "top-down" prefrontal cortical inhibition of amygdala activity controls emotional responses to social stimuli. A growing literature suggests that hypoactivity in the medial prefrontal cortex coupled with increases in amygdala activity underscore the vulnerability of CD individuals to relapse. Neuroimaging studies of corticolimbic network activity (functional connectivity) have been conducted in CD subjects at rest. Compared with healthy controls, CD subjects exhibited lower corticolimbic connectivity and the degree of corticolimbic uncoupling was associated with time to relapse. Studies measuring corticolimbic connectivity during exposure to a social stress task in CD subjects could provide critical insight into the neurobiologic mechanisms that underscore the sensitivity of CD individuals to social stress. Moreover interventions that improve corticolimbic connectivity in CD subjects may be effective therapeutic strategies for preventing relapse in CD populations. Oxytocin (OT) is an anxiolytic neuropeptide that attenuates amygdala responses to aversive social cues. In order to better understand the neurobiologic mechanisms that control emotion-related behavior in CD populations, we propose a double-blind placebo (PBO) controlled study using blood oxygen level dependent (BOLD) functional magnetic resonance imaging (fMRI) to measure (1) corticolimbic functional connectivity during the Montreal Imaging Stress Task (MIST) and (2) amygdala activity in response to an implicit facial affect recognition paradigm in groups of CD individuals (CD n=80) and healthy non-dependent controls (HC, n=80). Prior to the scanning session, participants will receive either intranasal OT (24 IU) or PBO spray (n=40 per treatment group). The order of the tasks will be counterbalanced.

DETAILED DESCRIPTION:
Individuals will be screened for eligibility over the telephone by a trained research assistant during which major inclusion/exclusion criteria will be assessed. Individuals who appear eligible will be invited for an in-person interview with a member of the research team. Prior to any study procedures, the individual will sign an Institutional Review Board (IRB) approved informed consent form. Following consent, a battery of standardized assessments will be delivered (described below). A general medical history and physical exam will also be performed to ensure that the subject is eligible to participate. The exam will also include a metal screening questionnaire that will be reviewed by clinical staff. If a patient is ineligible to participate, he or she will be given a referral for medical care and/or an appropriate treatment program.

C3e. Assessments Screening and Diagnostic Instruments Quick Screen: This assessment will quickly determine whether an individual meets study inclusion or exclusion criteria. The instrument is designed to assess for substance dependence and obvious psychiatric, medical, and logistic exclusions.

Mini-International Neuropsychiatric Interview (MINI): The MINI is a brief structured interview that was designed to assess Diagnostic and Statistical Manual (DSM) IV diagnoses using a series of questions in dichotomous format (yes/no). To date the MINI has not been revised to assess DSM V criteria. Earlier studies have found that the MINI is similar in sensitivity, specificity, and inter-rater reliability to other more lengthy diagnostic interviews, such as the SCID-I/P.

Structured Clinical Interview for DSM-IV (SCID-I/P): The SCID-P is a structured diagnostic interview that assesses each of the criteria for DSM-IV diagnoses. To date the SCID has not been revised to assess DSM-5 criteria. The alcohol and drug use disorder modules will be used to thoroughly assess both current and lifetime diagnostic status for abuse and dependence. It has excellent inter-rater and test-retest reliability.

Childhood Trauma Questionnaire (CTQ): Since childhood trauma has been shown to affect corticolimbic brain activity and corticolimbic brain activity following OT administration we will use the CTQ to assess childhood trauma exposure in each of the study participants. The CTQ is a 25-item self-report questionnaire used to assess the extent to which individuals have childhood abuse and neglect. Subjects answer each question using a 5-point Likert scale ranging from (1) never true to 5 (very often true). The reliability and validity of the CTQ have been tested in both healthy and substance-dependent populations.

Within Session Rating Scale: A modification of the Within Session Rating Scale will be used to assess craving and mood during the procedures. This scale is anchored with the adjectival modifiers ("not at all and extremely"). There are four items assessing domains of craving (want/need/craving/ability to resist). For the market value item, the individual will be asked to name the dollar amount they would be willing to pay for cocaine if they could have it "now". Other items include anxiety and mood. These data will be collected prior to treatment, prior to MIST1, and immediately after each run of the MIST.

Menstrual History Diary: Drug craving mood and affect have been associated with menstrual cycle phase and ovarian hormone status. Subjects will be asked to estimate the timing of their cycle for the 90-days prior to study entry and to track their cycle during study participation. Daily Hassles Scale: The Daily Hassles Scale consists of a list of 117 irritating, frustrating or distressing events that characterize everyday interactions with the environment. Subjects rate intensity for the past month. The Daily Hassles Scale is positively correlated with adaptational outcomes and is a good predictor of psychological symptoms. Data from the daily hassles will be used to explore the relationship between stress related corticolimbic brain activity and sensitivity to daily hassles.

Metal Screening Questionnaire (MSQ): The MSQ is a list of 18 "yes or no" questions regarding pacemakers, shrapnel, bullets, implants, tattoos, hairpieces, insulin pumps, cochlear implants, staples and metal clips, false eyes, nerve stimulators, dental bridges, replacement valves, intrauterine devices (IUDs), dentures, trans-dermal nicotine patches, surgery, metal in the eyes, claustrophobia, and current pregnancy. In addition the MSQ asks "have you ever been shot at or received treated for metal in your eyes?" The questionnaire is anchored by "Is there any possibility of metal, metal pieces, or metal implants in your body?" Each study participant will be asked to fill-out the MSQ at the assessment visit and the clinician will review the MSQ with the participant during the physical exam.

Minnesota Nicotine Withdrawal Scale (MNWS): Nicotine withdrawal could have a significant impact on our study outcomes. The MNWS is a 15-item self-report scale of behaviors associated with nicotine withdrawal. Subjects answer each question using a 5-point Likert scale ranging from (0) none to 4 (severe). Smokers will be asked to fill-out the questionnaire both before (prior to medication administration) and after the scanning sessions. Group differences in the severity of nicotine withdrawal may be used as covariates in the analysis.

The Connor-Davidson Resilience Scale (CD-RISC): The CD-RISC is a 25-item self-report measure that assesses the ability to cope with stress and adversity. Participants will be asked to complete the CD-RISC at the assessment visit.

Interpersonal Support Evaluation List Short Form (ISEL-SF): The ISEL-SF is a 12-item self-report form that measures perceived availability of four domains of social support (belonging, self-esteem, appraisal and tangible). Individuals rate each item using a four-point scale ranging from definitely false (1) to definitely true (4). Participants will be asked to complete the ISEL-SF at the assessment visit.

Urine Pregnancy Test: Female participants will be asked to provide a urine sample which will be tested for the presence of human chorionic gonadotropin (hCG) using the QuickVue One-Step urine hCG pregnancy test (Quidel Corporation, San Diego, CA). The test provides a qualitative measure of hCG in urine (≥ 25 milli-Intenational unit (mIU/mL); 99% sensitivity; 99% specificity). The urine pregnancy test will be performed at screening and on the day of the study visit, prior to the urine drug screen and breathalyzer test. If the pregnancy test is positive, the subject will be excluded and no further testing will take place.

Blood Sample Collection and Assays: Baseline saliva samples for estradiol, progesterone and a baseline blood sample for OT will be collected from each participant 15-30 minutes prior to the OT/PBO administration. Blood will be collected in tubes containing ethylenediaminetetraacetic acid (EDTA). Tubes will be centrifuged at 1500 rpm at 4˚C. Plasma will be stored at -70˚C. Determination of OT will be performed using a commercial ELISA kit (Enzo Life Sciences). Intra-assay coefficients of variation for OT average ~3-5% and inter-assay variation is typically less than 10%.

Substance Related Instruments Form 90: The Form 90, an assessment instrument commonly used in addiction studies, is similar in concept to the Time Line Follow back. This is a calendar-based instrument designed to assess daily substance consumption. Study participants will be asked to estimate the amount of substance consumed with the aid of visual cues designed to accurately quantify consumption. Cocaine will be recorded in dollar value as well as quantity in order to standardize for different types of cocaine use (crack, IV, nasal, etc.). The data will be summarized in three ways: (a) percent of abstinent days (i.e., no use); (b) amount of use per day and (c) days since last use.

Urine Drug Screening: Drug screens will be performed using the On Track Test Cup (Roche Diagnostics), an in vitro diagnostic test for the qualitative detection of drug or drug metabolite in the urine. The On Track Test Cup profile (cut off) consists of amphetamines (1000ng/ml), cocaine (300 ng/ml), tetrahydrocannabinol (THC) (50 ng/ml), morphine (300 ng/ml), and benzodiazepines (200 ng/ml). Results will be used to ascertain abstinence prior to initiation of test session and to substantiate self-report.

Breathalyzer: To ascertain abstinence from alcohol during the study period, subjects will have their breath sampled for the presence of alcohol (Alco-Sensor III, Intoximeters Inc., St. Louis, MO). The Alco-Sensor III can accurately detect breath alcohol levels between .000-.400 blood alcohol concentration (BAC).

Session Procedures Study Visit: Participants will be instructed to arrive at MUSC's Addiction Sciences Division (ASD) on the morning of the study visit. Participants will be informed that they will be expected to remain abstinent from cocaine and other drugs for the three-day period prior to the study visit in order to minimize the impact of recent drug/alcohol use on brain activity and subjective responses to the MIST. Participants will be asked to avoid caffeinated beverages on the morning of the study visit since caffeine may introduce variability in stress reactivity. If a participant is nicotine-dependent (s)he will be provided with a nicotine patch. Upon arriving at the ASD, the participant will be breathalyzed and will provide a urine sample, which will be tested for the presence of cocaine, opiates, barbiturates, benzodiazepines, and stimulants; if female, a urine pregnancy test will also be administered prior to the drug test. If the pregnancy and urine drug tests are negative,with the exception of marijuana, the session will proceed. In the event a participant tests positive for drugs or alcohol, the study visit will be rescheduled. Saliva samples will be collected, and the participant will be escorted to the Clinical Neurobiology Laboratory at the Institute of Psychiatry for a blood draw. Participants will then be escorted to the on-campus Center for Biomedical Imaging (CBI) facility by approved study personnel.

Medication Administration Intranasal OT and matching PBO (saline spray) will be compounded by MUSC's Investigational Drug Services (IDS) which has extensive experience in extemporaneous OT preparation and quality control monitoring. Randomization will be done by IDS, who will keep a record of the blind. The record will be available should unblinding be required. To achieve balance in sample size with respect to gender, smoking status, age, and race, a block randomized design with randomly varying block sizes will be used. OT or PBO sprays will be administered at the CBI and under the supervision of the study staff at 11:30 a.m., approximately 45-minutes prior to the scanning session. First the participant will be asked to blow their nose. The vial will be primed to ensure that each puff contains OT or placebo spray and not air. The participant will be instructed to exhale through their nose and then spray into one nostril while inhaling. Nostrils will be alternated and the participant will be asked to repeat the procedure for each nostril. Participants will self-administer three puffs of the nasal spray per nostril (4 IU of OT/puff) for a total of 24 IU. This dose and timing of administration were selected based on similar fMRI studies demonstrating BOLD signal changes in the amygdala 45-50 minutes post-administration.

MRI Data Acquisition All MRI data will be acquired on a Siemens Trio 3 Tesla (T) scanner (Siemens Medical, Erlangen, Germany). Participants will be screened for metal using a handheld metal detector. Study personnel will position subjects on the scanner bed with foam padding placed around their head to prevent motion. Participants will wear earplugs/headphones and the task will be projected on a wide screen located at the end of the scanner bore and viewed via a back-projected mirror that will be mounted on 12-channel head coil. Participants will use a non-ferrous optical hand pad to submit their answers to the arithmetic task. The hand pad will be connected via an optical cable to a computer outside the scanner room. Their ability to view the projection screen and use of the hand pad will be assessed prior to scanning. During initial scanner tuning, localizing, and structural scanning, participants will be shown "relaxing" images (i.e., 20 scenic pictures, each displayed for 30 seconds). A high resolution T1-weighted MPRAGE anatomical scan (TR = 8.1 ms, echo time (TE) (TE = 3.7 ms, flip angle = 8°, field of view = 256 mm, 1.0 mm) covering the entire brain and positioned using a sagittal scout image will be acquired for co-registration and normalization of functional images. T2*-weighted gradient echo planar imaging (EPI) images will be acquired with the following parameters: TR = 2500 ms, TE = 27 ms, flip angle = 77º, 40 axial slices (FOV = 224 x 224 mm, thickness = 3.5 mm voxels with 0.5 mm gap, in interleaved order. The scanning planes will be oriented parallel to the anterior commissure-posterior commissure line.

Implicit Facial Affect Recognition Task The amygdala response to emotional faces that are presented outside the focus of attention (i.e. implicit tasks) is significantly greater than that observed during overt (explicit) presentation of the same stimuli. Emotional adult faces will be selected from a variety of sources are standardized in size and enclosed in the same oval surround. Dr. Joseph (Co-I) has developed a corpus of faces for a recent project, "A comparative developmental connectivity study of face processing") that will be used for the present project. The faces will depict male and female Caucasian, Asian and African Americans expressing three different categories of emotion; fear, anger, and happiness. Neutral faces will also be presented. Because the participants will also be from different ethnic categories, it is important to include a mixture of races. In a block design, participants will view a series of faces (for 27.5 sec) within a block and report on the gender of those faces at the end of the block (for 5 sec). Each block will present 56 faces that depict the same emotion and same gender so there will be 6 pseudorandomly ordered task blocks (3 emotions x 2 genders) and 7 rest blocks (27.5 sec each) that present a crossbar to be fixated. In each task block, each emotional face will be presented for 33 msec. followed by a neutral face mask (from a different individual) for 167 msec. followed by a blank screen for 291 msec. At the end of the block participants will report the gender using two buttons on a response pad. Assignment of face sets to sessions will be counterbalanced across subjects.

The Montreal Imaging Stress Task The study will use a block design of three, six-minute runs separated by two-minutes of rest for feedback, for a total of 24-minutes. During each run, participants will be exposed to 40-second blocks of three different conditions (rest, control, and stress). Prior to the task, a research assistant will meet with each participant and described the parameters of the task. The participants will be shown images of what the screen will look like during each condition. The participants will be instructed to relax during the rest condition and focus on the screen. During the control condition, the participants will be asked to answer math problems as accurately as possible but will also be told that their responses will not be recorded. During the stress condition, the participants will be asked to perform the math task as quickly and accurately as possible. They will be given immediate feedback about their performance and will be able to see the performance level of an "average" person through a performance bar that will be located at the top of the screen. A strict time limit will be enforced throughout the stress condition. The participants will be told that the average person would answer about 85% of the questions correctly, while in reality, the program's algorithm limits the participants' performance rate to between 35-45%. At the end of runs one and two, the participants will be given negative feedback from the investigator and will be urged to improve their performance so that their data may be included in the study. To minimize the effects of scanner drift, the beginning condition will be counterbalanced between participants. However, the sequence of conditions will be constant (i.e. control condition will follow the rest condition and the stress condition will follow the control condition).

ELIGIBILITY:
General Inclusion/Exclusion Criteria Inclusion Criteria

1. Age 18-65.
2. Subjects must be able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.
3. Subjects must consent to remain abstinent from all drugs of abuse (except nicotine) for the three-day period immediately prior to the study visit.
4. Subjects must consent to random assignment.
5. Subjects must have a negative breathalyzer, urine drug screen at the study visit.
6. Subjects must consent to the study visit which includes an outpatient visit to the ASD and completing one functional magnetic resonance imaging (fMRI) scanning session.

Exclusion Criteria

1. Subjects with evidence of or a history of significant hematological, endocrine, cardiovascular, pulmonary, renal, gastrointestinal, or neurological disease including diabetes.
2. Subjects with a history of or current psychotic disorder or bipolar affective disorder.
3. Subjects with current major depressive disorder or post-traumatic stress disorder.
4. Subjects taking any psychotropic medications, including SSRI's or other antidepressants, opiates or opiate antagonists. Subjects taking trazodone or non-benzodiazepene hypnotics for sleep will be included.
5. Women who are pregnant, nursing or of childbearing potential and not practicing an effective means of birth control.
6. Subjects who have a BMI that procludes them from fitting comfortably in the scanner.
7. Persons with ferrous metal implants or pacemaker.
8. Subjects that are claustrophobic.
9. Subjects with significant psychiatric or medical problems that would impair participation or limit ability to complete the scanning session.
10. Subjects that require maintenance or acute treatment with any psychoactive medication including anti-seizure medications which could potentially interfere with fMRI data acquisition.

Group - Specific Inclusion/Exclusion Criteria Individuals with Cocaine Dependence Inclusion Criteria

1. Subjects must meet DSM-5 criteria for current (three months prior to study visit) moderate to severe cocaine use disorder. Individuals may meet criteria for mild marijuana use disorder, but they must not meet criteria for substance use disorder for any other substance (except nicotine) within the 60 days prior to study participation. Due to the high comorbidity of alcohol and cocaine use disorder individuals with alcohol use disorder will be included in the study if they do not require medically supervised detoxification.

Exclusion Criteria 1. Subjects meeting DSM-5 criteria for substance use disorder (other than nicotine, cocaine, marijuana or alcohol) within the 60 days prior to study participation.

Healthy Controls Inclusion Criteria

1. As above. Exclusion Criteria

1. Subjects meeting DSM-5 criteria for current or lifetime substance use disorder on any drugs of abuse (except nicotine and marijuana.
2. Subjects meeting DSM-5 criteria for marijuana use disorder within the last year.
3. Subjects with current major depression or post-traumatic stress disorder (past month)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2015-07; Primary Completion 2020-07-27 (Actual); Study Completion 2020-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee L McRae-Clark, PharmD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo/Cocaine User: Individuals who meet criteria for cocaine use disorder and are randomized to placebo.
  Placebo
- Placebo/Control: Healthy controls who are randomized to placebo.
  Placebo
Period: Overall Study
Arm/Group | Oxytocin/Cocaine User | Placebo/Cocaine User | Oxytocin/Control | Placebo/Control
Started | 40 | 37 | 29 | 32
Completed | 39 | 35 | 27 | 29
Not Completed | 1 | 2 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 2
Not completed — Physician Decision | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin/Cocaine User | Placebo/Cocaine User | Oxytocin/Control | Placebo/Control | Total
Number analyzed (Participants) | 39 | 35 | 27 | 29 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 39 | 34 | 27 | 29 | 129
  >=65 years | 0 | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 15 | 13 | 57
  Male | 26 | 19 | 12 | 16 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 39 | 35 | 26 | 28 | 128
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 39 | 35 | 27 | 29 | 130

OUTCOME MEASURES:

1. Primary Outcome: Functional Connectivity Between Corticolimbic Brain Regions During Acute Social Stress
Description: Psychophysiological interaction (PPI) analysis measures how strongly one region of the brain is connected to another brain region during a particular experimental condition, such as doing arithmetic while being given feedback about performance. The strength of this functional connection between two regions can be expressed as a parameter estimate - the higher the value of the parameter estimate, the more strongly connected the two regions are so that as activation in one region increases, activation in the connected region also increases. However, two regions can also be strongly negatively connected such that if activation in one region goes up during a task condition, activation in the other region goes down
Time Frame: During Montreal Imaging Stress Task in fMRI scanner
Population: Some scans were not useable to due to head movement.
Measure: Mean (Standard Deviation); unit: Arbitrary units
Arm/Group | Oxytocin/Cocaine User | Placebo/Cocaine User | Oxytocin/Control | Placebo/Control
Number analyzed (Participants) | 35 | 27 | 27 | 24
Arbitrary units | .011 (.099) | .012 (.103) | .043 (.097) | .0008 (.149)

2. Primary Outcome: Amygdala Activity in Response to Fearful Faces
Description: Use an implicit facial affect recognition paradigm to determine the impact of cocaine dependence and oxytocin on amygdala activity in response to fearful faces. The BOLD signal measured during neutral faces will be subtracted from the BOLD signal measured during fearful faces.
Time Frame: During Facial Recognition Task in fMRI scanner
Population: Some scans were not useable due to head movement.
Measure: Mean (Standard Deviation); unit: Bold signal
Arm/Group | Oxytocin/Cocaine User | Placebo/Cocaine User | Oxytocin/Control | Placebo/Control
Number analyzed (Participants) | 30 | 18 | 23 | 24
Bold signal | 8.33 (48.9) | 2.32 (47.6) | 11.98 (30.4) | 18.07 (30.8)

ADVERSE EVENTS:
Time Frame: Participants had one-time administration of oxytocin or placebo. Participants were monitored for 1.5 hours after administration.
Arm/Group | Oxytocin/Cocaine User | Placebo/Cocaine User | Oxytocin/Control | Placebo/Control
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/35 | 0/27 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/35 | 0/27 | 0/29
Other Adverse Events (participants affected / at risk) | 0/39 | 0/35 | 0/27 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT02682784/Prot_SAP_000.pdf